CLINICAL TRIAL: NCT04467073
Title: Examining a Stepped-care Telehealth Program for Parents of Young Children With Autism: a Proof of Concept Trial
Brief Title: Stepped-care Telehealth for Young Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Allison Wainer, Ph.D., Research Director, AARTS Center, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15100203
Record Dates: First submitted 2020-06-26; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-Care Online Reciprocal Imitation Training (Online RIT) (Experimental): Participants completed four telehealth modules over a period of 5 weeks (~1 per week, 1 week to practice). Two variables were selected as tailoring variables for this stepped-care model. Fidelity (RIT-PFF) and self-efficacy (EIPSES) at 5 weeks were used to determine which participants were in need of a "step up" in care, in the form of remote parent coaching.
  Parents who demonstrated ≥80% on the RIT-PFF, and who reported gains on the EIPSES continued to have access to Online RIT and practiced on their own for the next 5 weeks, but did not receive any remote coaching. Parents who demonstrated <80% fidelity on the RIT-PFF and/or who didn't report increases in the EIPSES were directed into coaching. Coaching involved videoconferences once per week (wks. 6-10) with a parent coach (PI), and followed the occupational performance coaching model. Sessions included review of successes and challenges, parent practice with feedback, problem solving, and planning.
  Interventions: Behavioral: Online RIT
- Wait List Control (No Intervention): Participants provided with information about available community resources after randomization. These participants were given the opportunity to engage in the stepped-care format of Online RIT after the post-intervention data collection time point; however their data was included exclusively in control group analyses.

INTERVENTIONS:
Behavioral: Online RIT — Online RIT presents RIT techniques in four sequential learning modules: (1) Setting Up For Success (2) Imitating your Child (3) Describing Play (4) Teaching Object Imitation. Each learning module includes an instructional video, quiz, interactive exercises, and at-home planning and reflection. The website also includes a video library, Frequently Asked Questions, downloadable visual aids, links to relevant external resources, and a customizable "dashboard" that allows users to track their individualized goals and the amount of time they have spent working on their goals (e.g., practice log).
  Arms: Stepped-Care Online Reciprocal Imitation Training (Online RIT)

SUMMARY:
This proof-of-concept study addresses the gap in the access to care literature by examining a stepped-care version of a telehealth naturalistic developmental behavioral intervention (NDBI), Online RIT. Online RIT is an interactive website introducing Reciprocal Imitation Training (RIT), an NDBI focused on enhancing social imitation. RIT uses a naturalistic behavioral approach to teach object and gesture imitation to young children with ASD within a play-based context. The efficacy of RIT has been demonstrated through a small randomized control trial, several single-subject design studies, as well as in independent replications. Prior research also suggests that parents can be taught to effectively use RIT with their children in person, and two single-subject design studies detail the development and feasibility testing of Online RIT plus therapist assistance. These preliminary data suggest Online RIT may serve as an ideal platform for examining the potential of individualized telehealth delivery formats, such as stepped-care. Therefore, the goal of this study was to compare a stepped-care format of Online RIT to a waitlist control condition to determine initial feasibility and effectiveness of this innovative intervention and service delivery model.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of ASD or significant concerns of ASD
* Parent reported imitation deficits

Exclusion Criteria:

* Children of parents who are non-English speaking
* Actively participating in other parent training programs

Ages: 16 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline RIT Parent Fidelity Form (RIT-PFF) Score at 15 weeks | Baseline and 15 weeks
  Trained observers scored the parent-child interactions for parent fidelity of the RIT intervention techniques.
Change from Baseline Unstructured Imitation Assessment (UIA) Score at 15 weeks | Baseline and 15 weeks
  The UIA was used to measure child social imitation. It is a standardized assessment that evaluates spontaneous imitation of actions with objects and gestures during play.
Change from Baseline Early Intervention Parenting Self-Efficacy Scale (EIPSES) Score at 15 weeks | Baseline and 15 weeks
  The EIPSES is a 20-item parent questionnaire designed to measure parenting efficacy within the context of early intervention.

SECONDARY OUTCOMES:
Change from Baseline Social Communication Checklist (SCC) Score at 15 weeks | Baseline and 15 weeks
  The SCC is a 47-item checklist completed by parents to indicate if a child uses a specific social communication skill.
Change from Baseline Beach Center Family Quality of Life Scale (FQOL) Score at 15 weeks | Baseline and 15 weeks
  The FQOL Scale is a 25-item self-report measure designed to assess family interaction, parenting, emotional well-being, physical/maternal well-being, and disability-related supports.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wainer AL, Arnold ZE, Leonczyk C, Valluripalli Soorya L. Examining a stepped-care telehealth program for parents of young children with autism: a proof-of-concept trial. Mol Autism. 2021 May 8;12(1):32. doi: 10.1186/s13229-021-00443-9. PMID 33964979